CLINICAL TRIAL: NCT01291173
Title: A Phase 2, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, Forced-dose Titration Study to Evaluate the Efficacy, Safety, and Tolerability of SPD489 in Adults Aged 18-55 Years With Binge Eating Disorder
Brief Title: Forced-dose Titration of SPD489 in Adults With Binge Eating Disorder
Acronym: BED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-208
Record Dates: First submitted 2011-02-04; First posted 2011-02-08 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SPD489 30 mg (Experimental)
  Interventions: Drug: lisdexamfetamine dimesylate (SPD489)
- SPD489 50 mg (Experimental)
  Interventions: Drug: lisdexamfetamine dimesylate (SPD489)
- SPD489 70 mg (Experimental)
  Interventions: Drug: lisdexamfetamine dimesylate (SPD489)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lisdexamfetamine dimesylate (SPD489) — SPD489-30mg capsules taken once daily for up to 11 weeks
  Other Names: LDX, Vyvanse
  Arms: SPD489 30 mg
Drug: lisdexamfetamine dimesylate (SPD489) — SPD489 50mg capsules taken once-daily for up to 11 weeks
  Other Names: LDX, Vyvanse
  Arms: SPD489 50 mg
Drug: lisdexamfetamine dimesylate (SPD489) — SPD489 70mg capsule taken once-daily for up to 11 weeks
  Other Names: LDX, Vyvanse
  Arms: SPD489 70 mg
Drug: Placebo — Placebo capsule taken once daily for up to 11 weeks
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of SPD489 compared to placebo in the treatment of moderate to severe binge eating disorder as measured by the number of binge days per week

ELIGIBILITY:
Inclusion

* Subject meets the following Diagnostic and Statistical Manual of Mental Disorders Fourth Edition - Text Revision (DSM-IV-TR) criteria for a diagnosis of binge eating disorder (BED).
* Binge eating disorder is of at least moderate severity in which subjects report at least 3 binge eating days per week.
* Subject has a body mass index (BMI) of >24 and <46.

Exclusion

* Subject has concurrent symptoms of bulimia nervosa or anorexia nervosa.
* Subject is considered a suicide risk or risk to harm others.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2011-05-10 (Actual); Primary Completion 2012-01-30 (Actual); Study Completion 2012-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (31):
- United States (31):
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Southwestern Research, Inc., Beverly Hills, California
  - Scripps Clinical Research Services, La Jolla, California
  - Pharmacology Research Institute, Newport Beach, California
  - PCSD - Feighner Research, San Diego, California
  - Florida Clinical Research, Bradenton, Florida
  - Gulfcoast Clinical Research, Fort Myers, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Atlanta Institute of Medicine and Research, Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Vince and Assoc. Research, Overland Park, Kansas
  - Clinical Trials Technology, Inc., Prairie Village, Kansas
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Marc Hertzman, MD, PC, Rockville, Maryland
  - McLean Hospital, Belmont, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - Unniversity of Minnesota, Minneapolis, Minnesota
  - Weight Disorders Washington University School of Medicine, Dept of Psychiatry, St Louis, Missouri
  - Robert Lynn Horne, MD, Las Vegas, Nevada
  - Richmond Behavioral Associates, Staten Island, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Neuropsychiatric Research Institute, Fargo, North Dakota
  - Community Research, Cincinnati, Ohio
  - Lindner City of Hope, Mason, Ohio
  - Weight Management Center, Medical University of South Carolina, Charleston, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Clinical Trials, Austin, Texas
  - Drug Development, Inc., Houston, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia

REFERENCES:
- [Derived] McElroy SL, Hudson JI, Mitchell JE, Wilfley D, Ferreira-Cornwell MC, Gao J, Wang J, Whitaker T, Jonas J, Gasior M. Efficacy and safety of lisdexamfetamine for treatment of adults with moderate to severe binge-eating disorder: a randomized clinical trial. JAMA Psychiatry. 2015 Mar;72(3):235-46. doi: 10.1001/jamapsychiatry.2014.2162. PMID 25587645

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A site with 11 enrolled subjects was excluded from study. An external investigation was initiated for reasons unrelated to the respective study. Lacking information on the purpose or scope of the investigation, it was deemed prudent to exclude data from subjects enrolled at site from the primary analyses of efficacy and safety.
Groups:
- Lisdexamfetamine Dimesylate (SPD489) 30 mg: SPD489-30mg capsules taken once daily for up to 11 weeks
- Lisdexamfetamine Dimesylate (SPD489) 50 mg: SPD489 50mg capsules taken once-daily for up to 11 weeks
- Lisdexamfetamine Dimesylate (SPD489) 70 mg: SPD489 70mg capsule taken once-daily for up to 11 weeks
Period: Overall Study
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Started | 64 | 66 | 65 | 65
Completed | 47 | 51 | 52 | 52
Not Completed | 17 | 15 | 13 | 13
Not completed — Adverse Event | 0 | 3 | 1 | 3
Not completed — Protocol Violation | 7 | 2 | 2 | 5
Not completed — Withdrawal by Subject | 6 | 4 | 4 | 2
Not completed — Lost to Follow-up | 4 | 6 | 3 | 2
Not completed — Unable to meet visit schedule | 0 | 0 | 1 | 0
Not completed — Lack of compliance | 0 | 0 | 0 | 1
Not completed — Subject was unblinded | 0 | 0 | 1 | 0
Not completed — Excluded therapy | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set defined as all randomized subjects who had taken at least 1 dose of investigational product and who had at least 1 follow-up safety assessment completed. One subject in the Placebo group did not have a post-baseline safety assessment and was excluded from the safety population (n=259).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg | Total
Number analyzed (Participants) | 63 | 66 | 65 | 65 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (10.30) | 38.4 (11.14) | 39.6 (9.32) | 38.6 (10.01) | 38.7 (10.17)
Age, Customized [Count of Participants; unit: Participants]
  18-39 years | 35 | 35 | 30 | 34 | 134
  40-55 years | 28 | 31 | 35 | 31 | 125
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 57 | 50 | 55 | 211
  Male | 14 | 9 | 15 | 10 | 48
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63 | 66 | 65 | 65 | 259

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Log Transformed Binge Days Per Week at Week 11
Description: Binge day is defined as a day during which at least 1 binge episode occurs.
Time Frame: Baseline and week 11
Population: Full Analysis Set defined as all subjects who had taken at least 1 dose of investigational product and who had 1 post-baseline primary efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: Log days
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Number analyzed (Participants) | 62 | 66 | 64 | 63
Log days | -1.23 (0.069) | -1.24 (0.067) | -1.49 (0.066) | -1.57 (0.067)
Statistical Analysis 1: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Test type: Superiority or Other; p = 0.8825, Mixed Models Analysis; Mean Difference (Final Values) = -0.014, 95% CI 2-sided [-0.203 to 0.175]
Statistical Analysis 2: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Test type: Superiority or Other; p = 0.0077, Mixed Models Analysis; Mean Difference (Final Values) = -0.258, 95% CI 2-sided [-0.446 to -0.069]
Statistical Analysis 3: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = -0.345, 95% CI 2-sided [-0.534 to -0.155]

2. Secondary Outcome: Change From Baseline in the Number of Binge Episodes Per Week at Up to 11 Weeks
Description: The number of binge episodes per week as assessed by clinical interview based on subject diary.
Time Frame: Baseline and up to 11 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Binge Episodes
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Number analyzed (Participants) | 62 | 66 | 64 | 63
Binge Episodes | -4.07 (2.718) | -4.57 (3.266) | -5.10 (3.026) | -5.09 (2.586)
Statistical Analysis 1: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Test type: Superiority or Other; p = 0.4676, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Test type: Superiority or Other; p = 0.0198, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Test type: Superiority or Other; p = 0.0031, Cochran-Mantel-Haenszel

3. Secondary Outcome: 1-Week Binge Response, Last Observation Carried Forward (LOCF)
Description: The 1-week binge response was defined as either a 1-week remission (a 100% reduction of binge episodes from baseline [ie, a cessation of binge eating behavior]), or a marked response (75 to <100% reduction in binge episodes from baseline), or a moderate response (50 to <75% reduction in binge episodes from baseline), or a negative/minimal response (<50% reduction in binge episodes from baseline). The 1-week response was determined at the end of the study utilizing a LOCF approach.
Time Frame: Last 7 days on study
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Number analyzed (Participants) | 62 | 66 | 64 | 63
Participants
  1 week remission | 23 | 28 | 33 | 35
  Marked response | 15 | 20 | 24 | 23
  Moderate response | 13 | 8 | 4 | 1
  Negative/Minimal response | 11 | 10 | 3 | 4
Statistical Analysis 1: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Test type: Superiority or Other; p = 0.3341, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Test type: Superiority or Other; p = 0.0063, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Test type: Superiority or Other; p = 0.0022, Cochran-Mantel-Haenszel

4. Secondary Outcome: 4-Week Binge Response
Description: Subjects are free from binge episodes for 4 weeks.
Time Frame: Last 28 days on study
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Number analyzed (Participants) | 61 | 63 | 64 | 62
Participants | 13 | 22 | 27 | 31
Statistical Analysis 1: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Test type: Superiority or Other; p = 0.0937, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Test type: Superiority or Other; p = 0.0127, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel

5. Secondary Outcome: Percent of Participants With Clinical Global Impression - Severity of Illness (CGI-S) at Baseline
Description: CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill)
Time Frame: Baseline
Population: Full Analysis Set defined as all subjects who had taken at least 1 dose of investigational product and who had 1 post-baseline primary efficacy assessment. (Not all subjects in the FAS had an assessment for this outcome.)
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Number analyzed (Participants) | 62 | 66 | 64 | 63
Percentage of participants
  Normal, not at all ill | 0 | 0 | 0 | 0
  Borderline mentally ill | 0 | 0 | 0 | 1.6
  Mildly ill | 1.6 | 0 | 3.1 | 1.6
  Moderately ill | 56.5 | 54.5 | 59.4 | 42.9
  Markedly ill | 29.0 | 30.3 | 29.7 | 47.6
  Severely ill | 11.3 | 12.1 | 6.3 | 6.3
  Among the most extremely ill | 1.6 | 3.0 | 1.6 | 0

6. Secondary Outcome: Percent of Participants With Clinical Global Impression - Severity of Illness (CGI-S) at Up to 11 Weeks
Description: as for outcome 5
Time Frame: up to 11 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Number analyzed (Participants) | 62 | 65 | 64 | 63
Percentage of participants
  Normal, not at all ill | 37.1 | 55.4 | 60.9 | 65.1
  Borderline mentally ill | 19.4 | 26.2 | 23.4 | 20.6
  Mildly ill | 12.9 | 1.5 | 6.3 | 11.1
  Moderately ill | 24.2 | 13.8 | 7.8 | 3.2
  Markedly ill | 6.5 | 1.5 | 1.6 | 0
  Severely ill | 0 | 0 | 0 | 0
  Among the most extremely ill | 0 | 1.5 | 0 | 0

7. Secondary Outcome: Percentage of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I) at Up to 11 Weeks
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: Up to 11 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Number analyzed (Participants) | 62 | 65 | 64 | 63
Percentage of participants | 64.5 | 84.6 | 90.6 | 93.7
Statistical Analysis 1: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Test type: Superiority or Other; p = 0.0091, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Test type: Superiority or Other; p = 0.0004, Chi-squared
Statistical Analysis 3: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Test type: Superiority or Other; p < 0.0001, Chi-squared

8. Secondary Outcome: Change From Baseline in Yale-Brown Obsessive Compulsive Scale Modified for Binge Eating (YBOCS-BE) Total Score at Week 11
Description: The YBOCS-BE measures the obsession of binge-eating thoughts and compulsiveness of binge-eating behaviors. The scale is a clinician-rated, 10-item scale, each item rated from 0 (no symptoms) to 4 (extreme symptoms). Total scores range from 0 to 40. A score of 0-7 is sub-clinical; 8-15 is mild; 16-23 is moderate; 24-31 is severe; and 32-40 is extreme.
Time Frame: Baseline and week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Number analyzed (Participants) | 62 | 66 | 64 | 63
units on a scale | -12.0 (0.87) | -15.0 (0.84) | -15.3 (0.83) | -17.0 (0.83)
Statistical Analysis 1: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Test type: Superiority or Other; p = 0.0142, Mixed Models Analysis; Mean Difference (Final Values) = -2.97, 95% CI 2-sided [-5.34 to -0.60]
Statistical Analysis 2: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Test type: Superiority or Other; p = 0.0075, Mixed Models Analysis; Mean Difference (Final Values) = -3.25, 95% CI 2-sided [-5.62 to -0.88]
Statistical Analysis 3: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -4.93, 95% CI 2-sided [-7.30 to -2.56]

9. Secondary Outcome: Change From Baseline in Montgomery-Ǻsberg Depression Rating Scale (MADRS) Score at Week 11
Description: MADRS is a validated, 10-item rating scale with each item being scored on a scale from 0-6 with a total score ranging from 0-60. Lower scores indicate a decreased severity of depression.
Time Frame: Baseline and week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Number analyzed (Participants) | 62 | 66 | 64 | 63
units on a scale | -1.7 (0.35) | -1.9 (0.34) | -1.3 (0.33) | -1.6 (0.33)
Statistical Analysis 1: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Test type: Superiority or Other; p = 0.7538, Mixed Models Analysis; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-1.11 to 0.80]
Statistical Analysis 2: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Test type: Superiority or Other; p = 0.3062, Mixed Models Analysis; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-0.45 to 1.44]
Statistical Analysis 3: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Test type: Superiority or Other; p = 0.7697, Mixed Models Analysis; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.81 to 1.09]

10. Secondary Outcome: Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Score at Week 11
Description: The HAM-A is a rating scale developed to quantify the severity of anxiety symptomatology. It consists of 14 items, each defined by a series of symptoms. Each item is rated on a 5-point scale, ranging from 0 (not present) to 4 (severe) with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity, and 25-30 moderate to severe, and 31-56 severe anxiety.
Time Frame: Baseline and week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Number analyzed (Participants) | 62 | 66 | 64 | 63
units on a scale | -1.5 (0.30) | -0.9 (0.29) | -1.1 (0.29) | -0.6 (0.29)
Statistical Analysis 1: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Test type: Superiority or Other; p = 0.2046, Mixed Models Analysis; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [-0.29 to 1.35]
Statistical Analysis 2: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Test type: Superiority or Other; p = 0.3348, Mixed Models Analysis; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-0.42 to 1.22]
Statistical Analysis 3: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Test type: Superiority or Other; p = 0.0505, Mixed Models Analysis; Mean Difference (Final Values) = 0.81, 95% CI 2-sided [-0.00 to 1.63]

11. Secondary Outcome: Change From Baseline in Eating Inventory Score at Week 11
Description: The Eating Inventory also known as the Three-Factor Eating Questionnaire is a 51-item self-reported questionnaire intended to assess 3 dimensions of eating behavior: cognitive restraint of eating, disinhibition, and hunger. Cognitive restraint of eating consists of 20 items, disinhibition consists of 16 items, and hunger consists of 15 items. Each item scores either 0 or 1 point for a total score of 0-20 for cognitive restraint of eating, 0-16 for disinhibition, and 0-15 for hunger. A higher score is better for cognitive restraint of eating and lower scores are better for disinhibition and hunger.
Time Frame: Baseline and week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Number analyzed (Participants) | 62 | 66 | 64 | 63
units on a scale
  Cognitive restraint of eating | 2.5 (0.65) | 4.4 (0.62) | 3.8 (0.61) | 4.3 (0.62)
  Disinhibition | -3.8 (0.58) | -5.6 (0.56) | -6.3 (0.55) | -7.2 (0.56)
  Hunger | -3.3 (0.58) | -5.3 (0.56) | -6.0 (0.55) | -7.8 (0.56)
Statistical Analysis 1: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Cognitive Restraint of Eating; Test type: Superiority or Other; p = 0.0371, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Cognitive Restraint of Eating; Test type: Superiority or Other; p = 0.1380, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Cognitive Restraint of Eating; Test type: Superiority or Other; p = 0.0459, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Disinhibition; Test type: Superiority or Other; p = 0.0278, Mixed Models Analysis
Statistical Analysis 5: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Disinhibition; Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis
Statistical Analysis 6: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Disinhibition; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 7: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Hunger; Test type: Superiority or Other; p = 0.0149, Mixed Models Analysis
Statistical Analysis 8: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Hunger; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis
Statistical Analysis 9: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Hunger; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

12. Secondary Outcome: Change From Baseline in Binge Eating Scale (BES) Score at Week 11
Description: The BES is a 16-item self-reported questionnaire that is designed to assess behavioral, affective, and attitudinal components of the subjective experience of binge eating. The items are summed, with possible scores ranging from 0 to 46. A score of 27 or higher indicates severe binge-eating problems, and a score of 17 or lower designates no binge-eating problems.
Time Frame: Baseline and week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Number analyzed (Participants) | 62 | 66 | 64 | 63
units on a scale | -12.2 (1.28) | -16.1 (1.25) | -17.6 (1.24) | -20.6 (1.24)
Statistical Analysis 1: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-7.44 to -0.38]
Statistical Analysis 2: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -5.4, 95% CI 2-sided [-8.95 to -1.94]
Statistical Analysis 3: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -8.5, 95% CI 2-sided [-11.99 to -4.92]

13. Secondary Outcome: Change From Baseline in Barratt Impulsiveness Scale (BIS-11) Total Score at Week 11
Description: The BIS-11 is a self-reported 30-item questionnaire that measures impulsiveness using a 4-point Likert scale (rarely/never = 1, occasionally = 2, often = 3, almost always/always = 4). A Total Impulsivity score is calculated by summing the scores for each item. Possible scores range from 30 - 120. Higher scores indicate increased impulsiveness.
Time Frame: Baseline and week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Number analyzed (Participants) | 62 | 66 | 64 | 63
units on a scale | -3.1 (1.09) | -5.8 (1.05) | -5.2 (1.05) | -6.9 (1.05)
Statistical Analysis 1: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Test type: Superiority or Other; p = 0.0824, Mixed Models Analysis; Mean Difference (Final Values) = -2.65, 95% CI 2-sided [-5.64 to 0.34]
Statistical Analysis 2: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Test type: Superiority or Other; p = 0.1725, Mixed Models Analysis; Mean Difference (Final Values) = -2.07, 95% CI 2-sided [-5.05 to 0.91]
Statistical Analysis 3: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Test type: Superiority or Other; p = 0.0148, Mixed Models Analysis; Mean Difference (Final Values) = -3.71, 95% CI 2-sided [-6.69 to -0.73]

14. Secondary Outcome: Change From Baseline in Short Form-12 Health Survey (SF-12) Score at Week 11
Description: The SF-12 is a 12-item self-report questionnaire that is a subset of the SF-36 Health Survey. The survey captures physical and mental health. There are 8 subscales. Four of the subscales has one-item each; the other 4 have two-items each. For each subscale, a mean value was first computed and transformed to a position on a scale ranging from 0-100 (Z-transformation). The aggregate total scores are then transformed into a mean value ranging from 0 (lowest level of health) to 100 (highest level of health).
Time Frame: Baseline and week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Number analyzed (Participants) | 62 | 66 | 64 | 63
units on a scale
  Aggregate Physical Score | 1.3 (0.78) | 2.6 (0.75) | 2.4 (0.74) | 3.9 (0.75)
  Aggregate Mental Score | 4.9 (1.03) | 5.0 (1.00) | 5.5 (0.99) | 4.9 (1.00)
Statistical Analysis 1: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Aggregate Physical Score; Test type: Superiority or Other; p = 0.2504, Mixed Models Analysis; Mean Difference (Final Values) = 1.25, 95% CI 2-sided [-0.89 to 3.38]
Statistical Analysis 2: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Aggregate Physical Score; Test type: Superiority or Other; p = 0.3090, Mixed Models Analysis; Mean Difference (Final Values) = 1.09, 95% CI 2-sided [-1.02 to 3.21]
Statistical Analysis 3: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Aggregate Physical Score; Test type: Superiority or Other; p = 0.0216, Mixed Models Analysis; Mean Difference (Final Values) = 2.50, 95% CI 2-sided [0.37 to 4.64]
Statistical Analysis 4: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 30 mg; Aggregate Mental Score; Test type: Superiority or Other; p = 0.9587, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-2.75 to 2.90]
Statistical Analysis 5: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 50 mg; Aggregate Mental Score; Test type: Superiority or Other; p = 0.6530, Mixed Models Analysis; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [-2.17 to 3.45]
Statistical Analysis 6: Comparison: Placebo vs Lisdexamfetamine Dimesylate (SPD489) 70 mg; Aggregate Mental Score; Test type: Superiority or Other; p = 0.9814, Mixed Models Analysis; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-2.79 to 2.86]

ADVERSE EVENTS:
Arm/Group | Placebo | Lisdexamfetamine Dimesylate (SPD489) 30 mg | Lisdexamfetamine Dimesylate (SPD489) 50 mg | Lisdexamfetamine Dimesylate (SPD489) 70 mg
Serious Adverse Events (participants affected / at risk) | 0/63 | 2/66 | 0/65 | 1/65
Other Adverse Events (participants affected / at risk) | 37/63 | 57/66 | 56/65 | 53/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | Lisdexamfetamine Dimesylate (SPD489) 30 mg (N=66) | Lisdexamfetamine Dimesylate (SPD489) 50 mg (N=65) | Lisdexamfetamine Dimesylate (SPD489) 70 mg (N=65)
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | Lisdexamfetamine Dimesylate (SPD489) 30 mg (N=66) | Lisdexamfetamine Dimesylate (SPD489) 50 mg (N=65) | Lisdexamfetamine Dimesylate (SPD489) 70 mg (N=65)
Dry mouth (Gastrointestinal disorders) | 5 | 22 | 22 | 27
Decreased appetite (Metabolism and nutrition disorders) | 4 | 17 | 13 | 12
Insomnia (Psychiatric disorders) | 1 | 7 | 10 | 9
Headache (Nervous system disorders) | 6 | 9 | 9 | 5
Nausea (Gastrointestinal disorders) | 0 | 5 | 6 | 4
Constipation (Gastrointestinal disorders) | 1 | 6 | 3 | 5
Nasopharyngitis (Infections and infestations) | 2 | 8 | 1 | 3
Weight decreased (Investigations) | 1 | 2 | 4 | 6
Irritability (General disorders) | 4 | 5 | 3 | 3
Diarrhea (Gastrointestinal disorders) | 0 | 4 | 5 | 1
Anxiety (Psychiatric disorders) | 0 | 4 | 4 | 1
Feeling jittery (General disorders) | 0 | 1 | 3 | 5
Palpitations (Cardiac disorders) | 0 | 4 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 3 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 3 | 3 | 2
Sleep disorder (Psychiatric disorders) | 0 | 1 | 3 | 4
Fatigue (General disorders) | 2 | 2 | 3 | 2
Initial insomnia (Psychiatric disorders) | 0 | 2 | 2 | 3
Energy increased (General disorders) | 0 | 2 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
External investigation at a site was initiated for reasons unrelated to the study. Lacking information on the investigation, it was deemed prudent to exclude data from subjects enrolled at site (n=11) from the primary analyses of efficacy and safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.